CLINICAL TRIAL: NCT05364580
Title: A Multicenter, Double-blind, Randomized, Parallel, Active-controlled, Phase III Clinical Trial to Compare the Efficacy and Safety of Protoxin Versus Botox® in Subjects With Moderate to Severe Glabellar Lines
Brief Title: The Efficacy and Safety Study of Protoxin Versus Botox® in Subjects With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protox Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT_BTA_P3_21
Record Dates: First submitted 2022-04-19; First posted 2022-05-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-03

CONDITIONS: Glabellar Frown Lines
Keywords: Glabellar Lines; Botulinum toxin; Botulinum toxin type A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROTOXIN(Phase Ⅲ) (Experimental): PROTOXIN will be injected to 5 glabellar lines (Each 4U/0.1mL, Total 20U/0.5mL)
  Interventions: Biological: PROTOXIN
- Botox® (Phase Ⅲ) (Active Comparator): Botox® will be injected to 5 glabellar lines (Each 4U/0.1mL, Total 20U/0.5mL).
  Interventions: Biological: Botox®

INTERVENTIONS:
Biological: PROTOXIN — Botulinum toxin Type A
  Arms: PROTOXIN(Phase Ⅲ)
Biological: Botox® — Botulinum toxin Type A
  Arms: Botox® (Phase Ⅲ)

SUMMARY:
This study will be conducted in Phase Ⅲ clinical trials. In Phase Ⅲ, subjects with moderate to severe glabellar lines are enrolled and those who are judged to be eligible for this study will be injected with the "PROTOXIN" at a total of 20U(4U/0.1mL each) in five sites of the glabellar lines. The investigational product is administered once, maintaining double-blind for a total of 16 weeks of observation. Thereafter, efficacy and safety are assessed by comparing with BOTOX® after regular visits conducted at 4,8,12 and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 19 to 65 years old
* Subjects attaining ≥grade 2 (moderate) in the investigator's rating of the severity of glabella lines at maximum frown
* Those who understand and comply with clinical trial procedures and visit schedules
* Subjects who voluntarily decides to participate and signs the consent form after hearing the explanation of this clinical trial.

Exclusion Criteria

* Those with or accompanied by the following diseases at the time of screening

  1. Subjects with Neuromuscular Junction Disorder that may affect neuromuscular action
  2. Subjects with previous history of weakness or paralysis in the forehead area
  3. Subjects with infection, skin disorders, or scars at the glabellar region
* Subjects with wrinkles that physically prevent wrinkles from spreading, such as when wrinkles are not spread out by hand
* Subjects who is administering a drug with muscle relaxation within four weeks of screening.
* Subjects who have taken Aspirin and NSAIDs within 7 days prior to administration of the investigational drug
* Subjects with surgical history who may affect wrinkles around the forehead or glabellar region
* Subjects who have planned facial cosmetic procedure during the clinical trial
* Subjects who have been administered similar drugs within 12 weeks (Botulinum toxin type A) or within 16 weeks (Botulinum toxin type B) before screening
* Subjects who are expected to administer botulinum toxin preparations other than Investigational product during the clinical trial period
* Subjects with allergy or hypersensitivity to the botulinum toxin or their components
* A history of drug or alcohol abuse
* Anxiety disorders or other significant mental disorders based on the judgment of an investigator
* Fertile women and men who have plans to conceive during pregnancy, breastfeeding and clinical trials or who do not agree to appropriate contraception
* Pregnant or lactating women
* Subjects with severe comorbidities or acute diseases that does not suitable for participation in clinical trials
* Those who participated in other clinical trials/clinical medical device trials within 30 days prior to screening and who received Investigational product/medical devices/procedures, or those who had less than 5 times the half-life of the Investigational product
* Subjects who are not eligible for this study based on the judgment of an investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving at least a 2-grade improvement from baseline on the facial wrinkle scale of GL at maximum frown at Week 4 | 4 weeks post injection compared to baseline
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe

SECONDARY OUTCOMES:
Investigator-rated improvement rate of glabellar lines at maximum frown | Week 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe
Participant-rated improvement rate of glabellar lines at maximum frown | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe
Investigator-rated improvement rate of glabellar lines at rest | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe
Participant-rated improvement rate of glabellar lines at rest | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe
Independent photo evaluator-rated improvement rate of glabellar lines at frown | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe
Independent photo evaluator-rated improvement rate of glabellar lines at rest | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe
Participant-rated satisfaction after treatment | Week 4, 8, 12, 16
  Participant evaluate the level of satisfaction by Patient Satisfaction(PS) 7-grade score(1 to 7) where 1 = very dissatisfied and 7 = very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Kim Beomjoon, Principal Investigator — Chung-Ang University Hospital, Chung-Ang University College of Medicine; Lee Yangwon, Principal Investigator — Konkuk University Medical Center; Kim Moonbeom, Principal Investigator — Pusan National University Hospital; Lee Jonghoon, Principal Investigator — Nown Eulji Medical Center, Eulji University; Shin Minkyung, Principal Investigator — Kyunghee University Medical Center
Locations (5):
- South Korea (5):
  - Kyung Hee University Hospital, Seoul, Dongdaemun-gu
  - Chung-Ang University Hospital, Seoul, Gwangjin-gu
  - Konkuk University Hospital, Seoul, Gwangjin-gu
  - Nowon Eulji Medical Center, Seoul, Nowon-gu
  - Pusan National University Hospital, Pusan, Seo-gu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Son HS, Shin MK, Lee JH, Kim MB, Yoo KH, Choi SY, Han HS, Seok J, Kim BJ, Lee YW. Efficacy and Safety of Novel Botulinum Toxin Type A (Protoxin) in the Treatment of Moderate to Severe Glabellar Lines: A Multicenter, Randomized, Double-Blind, Active-Controlled Phase III Study. Ann Dermatol. 2026 Feb;38(1):33-41. doi: 10.5021/ad.25.124. PMID 41607140